CLINICAL TRIAL: NCT02786797
Title: Efficacy of MBSR Treatment of Cognitive Impairment Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01CA199160-01 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-06-01 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; mindfulness-based stress reduction; cognitive impairment
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MBSR(BC) 6 Week Program (Experimental): Participants who are randomized to MBSR(BC) program will receive of educational material; group practice of mindfulness meditation (MM) and homework assignments; and group processes related to the practice of MM and supportive group interaction. Participants who receive MBSR will receive training in (1) sitting meditation anchored to the breath; (2) body scan (observing body sensations from the toes to the head); (3) Gentle Yoga (postures and stretches that increase awareness and balance; and (4) walking meditation. Through this arm of the study the goal is to enhance executive cognition through training in self-regulation of attention and acceptance of experience.
  Interventions: Behavioral: MBSR(BC) 6 Week Program
- BCES Education Support Program (Active Comparator): Participants who are randomized to the BCES program will be scheduled for 6 weekly, 2-hour sessions. BCES compared to MBSR(BC) meets the following criteria: (1) professional contact and group support time matched equally to the MBSR(BC) program; and (2) the content or activities of the BCES program does not include meditation or attention, relaxation, yoga, body scan, or walking meditation. This program is as an active control condition that accounts for nonspecific effects related to attention from the leader and favorable outcome expectancy, the educational materials provided and supportive interaction between group members and is matched for homework activity time over the 6 months. This group will be offered the MBSR(BC) program within 4 to 6 months after study completion.
  Interventions: Behavioral: BCES 6 Week Program
- Usual Care (No Intervention): Participants who are randomized to the Usual Care (UC) or control group will continue to receive standard post-treatment medical and nursing clinic visits that will not be modified by study participation. The UC participants will participate in their standard care appointments and will not be required to alter their UC regimen; however, they will be asked not to initiate a mindfulness program during the study period. The UC group will be offered the MBSR(BC) program within 4 to 6 months after study completion.

INTERVENTIONS:
Behavioral: MBSR(BC) 6 Week Program — The MBSR(BC) is a clinical program that provides systematic training to promote stress reduction by self-regulating arousal to stress. The goal of training is to teach participants to become more aware of their thoughts and feelings, and through meditation practice, to have the ability to step back from thoughts and feelings during stressful situations that contribute to increased emotional distress. It incorporates simple yoga, sitting meditation, body scan, and walking meditation in this program. Classes for this intervention occur on a weekly basis for 2 hours for 6 weeks. The participants will be asked to record their informal/formal practices in a daily diary during the program and from 6 weeks to 6 months after the intervention.
  Arms: MBSR(BC) 6 Week Program
Behavioral: BCES 6 Week Program — The BCES is an education support program. This 6-week program is based on the published NIH program, "Support for People with Cancer: Taking Time Education Support Group." In addition the class sessions consist of group discussion of educational materials and homework assignments; and group processes related to sharing supportive care situations. The participants will record their feelings, coping mechanisms, and questions related to survivorship in a daily diary during the program and from 6 weeks to 6 months after the intervention.
  Arms: BCES Education Support Program

SUMMARY:
The purpose of this study is to evaluate MBSR(BC), an intensive meditation-based stress reduction intervention, in order to determine its efficacy in improving cognitive functioning among breast cancer survivors. The study will employ a three group randomized design that will (1) evaluate the extent to which MBSR(BC) compared to the Breast Cancer-Education Support (BCES) program or Usual Care (UC) improves cognitive functioning among breast cancer survivors off treatment; (2) determine if improvements in cognitive functioning achieved from MBSR(BC) are mediated through increased mindfulness and decreased rumination and stress; (3) evaluate genetic variants as moderators of MBSR(BC) on improvements in CI; and (4) determine the impact of MBSR(BC) on healthcare utilization and costs, in addition it will be delivered to a sub-group in Spanish. If shown to be efficacious, the possibility exists of utilizing this intervention in other types of cancers as well as non-cancer health-related disorders in order to minimize the morbidity experienced by these populations.

DETAILED DESCRIPTION:
Due to improved detection and treatment, survival rates among breast cancer survivors have increased. However, breast cancer survivors may experience cognitive impairment (CI) following treatment, which has been reported by breast cancer survivors up to 10 years after chemotherapy (CT). There is limited evidence on whether stress-reducing interventions improve CI in breast cancer survivors. The primary goal of this application is to establish the Mindfulness-Based Stress Reduction for Breast Cancer (MBSR(BC)) program as an effective treatment for CI in breast cancer survivors. Specifically this study aim to (1) evaluate the extent to which MBSR(BC) compared to the Breast Cancer-Education Support (BCES) program or Usual Care (UC) improves cognitive functioning among breast cancer survivors off treatment; (2) determine if improvements in cognitive functioning achieved from MBSR(BC) are mediated through increased mindfulness and decreased rumination and stress; (3) evaluate genetic variants as moderators of MBSR(BC) on improvements in CI; and (4) determine the impact of MBSR(BC) on healthcare utilization and costs.

To achieve these aims, the research team will conduct a randomized controlled trial (RCT) among 300 breast cancer survivors (with an expected completed sample size of 250) with Stage I-III BC who have received adjuvant CT or CT and radiation. Within this RCT, MBSR(BC) will be delivered to a sub-population of Spanish speaking breast cancer survivors. Participants will be randomly assigned in a 1:1:1 ratio to 1 of 3 conditions (1) the 6-week MBSR(BC) program; (2) the 6-week BCES program; or (3) UC. However, once the UC condition has reached a total of 30 participants, then randomization at the baseline assessment will occur in a 1:1 ratio to 1 of 2 conditions: (1) MBSR(BC) and (2) BCES.

The BCES program will match the MBSR(BC) program for time and attention and parallel the group support component of MBSR(BC). Assessments will take place at baseline, 6 weeks,12 weeks and 6 months and include clinical history and demographic information, objective neuropsychological assessments, subjective cognitive and symptom measurements, cost utilization surveys, and either the blood or buccal (cheek) cells collection for genetic analyses.

This study is highly innovative to be the first randomized trial to: 1) evaluate the efficacy of MBSR(BC) among breast cancer survivors for objective neuropsychological and subjective improvements in cognitive functioning; 2) evaluate genetic profiles as moderators of MBSR(BC) on improving CI; 3) offer the MBSR trial in Spanish in addition to English for the purpose of improving cognition; and 4) determine the effect of MBSR(BC) on CT-induced CI among breast cancer survivors related to health service utilization costs.

MBSR(BC) provides training to promote stress reduction through self-regulation of attention and awareness to stressful events. The preliminary results show that MBSR(BC) improves subjective cognitive functioning. If MBSR(BC) is found to be effective, it will provide evidence of a viable non-pharmacological method for managing CI in breast cancer survivors. Additionally, the examination of the effects of the hypothesized mediators may yield new insights for tailoring MBSR(BC) and/or developing additional interventions to aid breast cancer survivors. The assessment of genetic polymorphisms to explore if risk alleles are associated with improvement in cognitive functioning may demonstrate that specific genetic profiles may modify improvements in CI for those receiving MBSR(BC). Finally, if MBSR(BC) is shown to be effective, this may significantly impact healthcare utilization and cost and produce necessary evidence for clinicians, researchers and policymakers.

ELIGIBILITY:
Inclusion Criteria:

* Women age 21 or older who have:

  1. a diagnosis of stage I, II, or III breast cancer;
  2. completed CT or CT and radiation and are within 5 years post-treatment;
  3. BC patients with a previous history of another cancer who have NOT received any chemotherapy or chemotherapy and radiation, but have only received surgical treatments are eligible;
  4. met the screening criteria for CI through a positive response to at least 1 of 2 scaled questions from the European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC-QLQ) i.e. Please rate on a scale from 0 to 10, the difficulty level you have in concentrating on things, like reading a newspaper or watching television? "0" means no difficulty and "10" means very difficult. Please rate on a scale from 0 to 10, the difficulty level you have in remembering things. "0" means no difficulty and "10" means very difficult, will be included.
  5. Subjects must have the ability to read and speak English and Spanish at the 8th grade level or above, and survivors with mild depression, anxiety, or other psychiatric conditions will be eligible.

     Exclusion Criteria:
* Breast cancer survivors with a severe current psychiatric diagnosis (e.g. bipolar disorder)
* Stage 0 or Stage IV BC
* History of another primary cancer diagnosis, treated with adjuvant chemotherapy
* Previous chemotherapy
* Current diagnosed neurologic disorder
* Or a traumatic brain injury will be excluded

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in Executive Functioning from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Executive functioning is assessing the ability to develop, carry out, and make necessary changes to plans that have a goal.
  This will be measured using the Stroop Neuropsychological Screening Test (SNST).

SECONDARY OUTCOMES:
Change in Executive Function from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Executive functioning is assessing the ability the ability to develop, carry out, and make necessary changes to plans that have a goal.
  This will be measured using the Color Trails Test (CTT-2) and the Symbol Digit Modalities Test (SDMT).
Change in Visuospatial Memory from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Visuospatial Memory is assessing the ability to see an object or a picture then reproduce the same object or picture if given in different parts.
  These will be measured using the Brief Visuospatial Memory Test-Revised (BVMT-R).
Change in Verbal Memory from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Verbal Memory is assessing the ability to listen to words then reproduce the words into categories if given in different parts.
  These will be measured using the Verbal Memory ( Hopkins Verbal Learning Test-Revised (HVLT-R).
Change in Logical Memory from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Logical Memory is assessing the ability to listen to a detailed story then reproduce the detailed story.
  These will be measured using the Logical memory (Logical Memory I sub-scales from the Wechsler Memory Scale-IV (WMS-IV).
Change in Attention and Concentration from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Attention and Concentration are assessing the ability to follow instructions and complete tasks given the specific or non-specific nature of these tasks.
  These will be measured using the Digit Span sub-test of the Wechsler Adult Intelligence Scale-IV and Part 1 of the Color Trails Test (CTT-1).
Change in Verbal fluency from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  Verbal fluency is assessing the ability to say as many words as possible from a category in a given time.
  This will be measured using the Controlled Oral Word Association Test (COWAT).
Change in Cognitive Functioning from baseline to 6 months. | Baseline, 6 weeks (post intervention), 12 weeks follow-up and 6 months follow-up.
  This will be measured using the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - USF Health Carol and Frank Morsani Center, Tampa, Florida
  - Florida Hospital Tampa, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lengacher CA, Hueluer G, Wang JR, Reich RR, Meng H, Park JY, Kip KE, Morgan S, Joshi A, Tinsley S, Krothapalli M, Nidamanur S, Cox C, Kiluk J, Lucas JM, Fonseca T, Moscoso MS, Bornstein E, Donovan KA, Padgett LS, Chamkeri R, Patel D, Hornback E, Rodriguez CCS. A Randomized Clinical Trial of Mindfulness-Based Stress Reduction Program Among Breast Cancer Survivors Post-Treatment: Evaluating Mediators of Cognitive Improvement. J Integr Complement Med. 2025 Apr;31(4):367-377. doi: 10.1089/jicm.2024.0493. Epub 2024 Dec 23. PMID 39711191
- [Derived] Park JY, Lengacher CA, Rodriguez CS, Meng H, Kip KE, Morgan S, Joshi A, Hueluer G, Wang JR, Tinsley S, Cox C, Kiluk J, Donovan KA, Moscoso M, Bornstein E, Lucas JM, Fonseca T, Krothapalli M, Padgett LS, Nidamanur S, Hornback E, Patel D, Chamkeri R, Reich RR. The Moderating Role of Genetics on the Effectiveness of the Mindfulness-Based Stress Reduction for Breast Cancer (MBSR(BC)) Program on Cognitive Impairment. Biol Res Nurs. 2025 Apr;27(2):216-228. doi: 10.1177/10998004241289629. Epub 2024 Oct 16. PMID 39413359
- [Derived] Lengacher CA, Reich RR, Rodriguez CS, Nguyen AT, Park JY, Meng H, Tinsley S, Hueluer G, Donovan KA, Moscoso MS, Bornstein E, Kiluk J, Nidamanur S, Padgett LS, Lucas JM, Fonseca T, Joshi A, Lin KJ, Goodman M, Kip KE. Efficacy of Mindfulness-Based Stress Reduction for Breast Cancer (MBSR(BC)) a Treatment for Cancer-related Cognitive Impairment (CRCI): A Randomized Controlled Trial. J Integr Complement Med. 2025 Jan;31(1):75-91. doi: 10.1089/jicm.2024.0184. Epub 2024 Sep 18. PMID 39291332
- See also: The 6-week curriculum is based on the published NIH program, "Support for People with Cancer: Taking Time Education Support Group." — https://www.cancer.gov/publications/patient-education/takingtime.pdf